CLINICAL TRIAL: NCT01841931
Title: Buprenorphine Tx:A Safe Alternative for Opioid Dependent Pain Patients
Brief Title: Buprenorphine Treatment: A Safe Alternative for Opioid Dependent Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is no longer at this site
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/09/VA05
Record Dates: First submitted 2013-01-25; First posted 2013-04-29 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2013-07

CONDITIONS: Opioid Use Disorder
Keywords: Opioids; Dependence; Buprenorphine; Pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Sublingual buprenorphine/naloxone taken in a 3 day induction, with a final daily dose (up to 32 mg depending on the subject) taken daily, as prescribed by the study psychiatrist. Subjects will continue buprenorphine for study duration (6 months).
  Other Names: Buprenorphine; Suboxone

SUMMARY:
The purpose of this study is to examine whether buprenorphine can be at least as effective as other opioid medications in relieving chronic pain in patients who suffer from dependence on their opioid medications, while patients simultaneously experience progressive decline of pain along with absence of opioid withdrawal symptoms and improved quality of life.

DETAILED DESCRIPTION:
The study will utilize sublingual buprenorphine for the treatment of chronic pain patients with co-occurring opioid dependence. Adult male and female chronic pain patients with co-occurring opioid dependence/disorder, being treated at MMC will be enrolled in a home induction procedure. Subjects will be switched from their current opioid pain medication to buprenorphine/naloxone to assess whether buprenorphine is at least as effective, if not more effective, as other opioid medications in controlling their pain while simultaneously improving their psychological distress, functional status, and other aspects of patients' lives. We will utilize a home induction procedure, and maintain subjects on this oral medication for a duration of 6 months. During this period

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM criteria for opioid dependence (or opioid use disorder when DSM 5 is in use)
* Has received opioid therapy for at least 90 days
* Has opioid dependence as assessed by a Maimonides psychiatrist

Exclusion Criteria:

* Scheduled for major surgery during study duration
* Predicted life expectancy < 1 year
* Plan to cease habitation in greater New York area within 6 months
* Risks for buprenorphine outweigh potential benefit, as determined by the PI
* Lacks sufficient fluency in English to understand the study protocol, answer survey questions or give informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kolodny, MD, Principal Investigator — Maimonides Medical Center Dept. of Psychiatry Chairman
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] TEDS. Treatment Episode Data Set, 1998-2008. Subsance Abuse and Mental Health Services Administration, Office of Applied Studies, http://wwwdasis.samhsa.gov/webt/NewMapv1.htm
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Walsh SL, Preston KL, Stitzer ML, Cone EJ, Bigelow GE. Clinical pharmacology of buprenorphine: ceiling effects at high doses. Clin Pharmacol Ther. 1994 May;55(5):569-80. doi: 10.1038/clpt.1994.71. PMID 8181201
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Rosen CS, Drescher KD, Moos RH, Finney JW, Murphy RT, Gusman F. Six- and ten-item indexes of psychological distress based on the Symptom Checklist-90. Assessment. 2000 Jun;7(2):103-11. doi: 10.1177/107319110000700201. PMID 10868247
- [Background] Sobell, L.C., & Sobell, M.B., Alcohol Timeline Followback (TFLB), in Handbook or Psychiatric Measures, I.A.P.A. (ed.), Editor. 2000, American Psychiatric Association: Washington, D.C. p. 477-479.
- [Background] Lee JD, Grossman E, DiRocco D, Gourevitch MN. Home buprenorphine/naloxone induction in primary care. J Gen Intern Med. 2009 Feb;24(2):226-32. doi: 10.1007/s11606-008-0866-8. Epub 2008 Dec 17. PMID 19089508
- [Background] Schilthuizen M, Stouthamer R. Horizontal transmission of parthenogenesis-inducing microbes in Trichogramma wasps. Proc Biol Sci. 1997 Mar 22;264(1380):361-6. doi: 10.1098/rspb.1997.0052. PMID 9107051
- See also: British Pain Society guidelines on prescribing opioids, intended for both doctors and patients. — http://www.britishpainsociety.org/book_opioid_main.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient: Enrolled patients
Period: Overall Study
Arm/Group | Patient
Started | 4
Completed | 0 (As the PI left the institution the study was terminated)
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Chronic pain patients with opioid dependence
Arm/Group | Patient
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Pain severity [Mean (Full Range); unit: units on a scale] — Pain Severity measured with a numeric scale (0 to 10) - Brief Pain Inventory (BPI)
  units on a scale | 7 [4 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Opiate Withdrawal
Description: Goal that patients will have NO withdrawal symptoms by the completion of their 3-day buprenorphine induction, and will remain withdrawal-free for the entire study duration.Assessed using Clinical Opiate Withdrawal Scale (COWS).
Time Frame: 6 months
Arm/Group | Patient
Number analyzed (Participants) | 0

2. Primary Outcome: Pain Severity
Description: Pain severity will be measured using a numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine), adopted from the Brief Pain Inventory (BPI).
  No results to report.
Time Frame: 6 months
Population: Enrolled patients
Arm/Group | Patient
Number analyzed (Participants) | 0

3. Secondary Outcome: Psychiatric Distress
Description: The investigators will utilize the SCL-6 (Symptoms Checklist 6, a validated abbreviated version of the SCL-90) to assess patients' psychological well being.
Time Frame: 6 months
Population: Enrolled patients
Arm/Group | Patient
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life
Description: Investigators will use the QOL (EuroQol EQ5D) questionnaire, which assess patients' self-assessment of health and health-related quality of life.
Time Frame: 6 months
Population: Enrolled patients
Arm/Group | Patient
Number analyzed (Participants) | 0

5. Secondary Outcome: Positive Affect
Description: The investigators will assess patients' moods/affects using the PANAS (Positive Affect Negative Affect Scale).
Time Frame: 6 months
Population: Enrolled patients
Arm/Group | Patient
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Patient
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Study was prematurely terminated as the PI left the institution.

Early termination lead to small numbers of subject enrollment and only baseline data. No data collection at 6 months or thereafter.

No adverse events.

No results to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes